CLINICAL TRIAL: NCT03728959
Title: Effects of a Liquid Meal and Gut Hormones (GIP and GLP-2) on Bone Remodeling in Participants With Hypoparathyroidism (KS-4-HypoPT).
Brief Title: Effects of a Liquid Meal and Gut Hormones (GIP and GLP-2) on Bone Remodeling in Participants With Hypoparathyroidism.
Acronym: KS-4-HypoPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, principal investigator. Cand.pharm., ph.d. student, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KS-4-HypoPT
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hypoparathyroidism
Keywords: hypoparathyroidism; Glucose-dependent insulinotropic polypeptide (GIP); Glucagon-like peptide-2 (GLP-2); Bone remodeling; Bone resorption; Bone formation; C-terminal telopeptide (CTX); N-terminal propeptide of type 1 procollagen (P1NP)
MeSH Terms: conditions — Hypoparathyroidism; Bone Resorption; Xanthomatosis, Cerebrotendinous | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Liquid meal (Nutridrink) (Experimental): Liquid meal (Nutridrink)
  Interventions: Other: Liquid meal (Nutridrink)
- GIP (Experimental): Glucose-dependent insulinotropic polypeptide
  Interventions: Other: GIP
- GLP-2 (Experimental): Glucagon-like peptide-2
  Interventions: Other: GLP-2
- Placebo (saline) (Experimental): Placebo (saline)
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Other: Liquid meal (Nutridrink) — Liquid meal ingested over 1 minute.
  Arms: Liquid meal (Nutridrink)
Other: GIP — Subcutaneous injected GIP
  Arms: GIP
Other: GLP-2 — Subcutaneous injected GLP-2
  Arms: GLP-2
Other: Placebo (saline) — Subcutaneous injected Placebo (saline)
  Arms: Placebo (saline)

SUMMARY:
Hypoparathyroidism (hypoPT) is characterized by low levels of PTH.

In this study we will test the effects of a liquid meal on the bone remodeling in participants with hypoparathyroidism. Furthermore, we will test the effects of the gut hormones GIP and GLP-2.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 76
* Hypoparathyroidism

Exclusion Criteria:

* Diabetes
* Disease in the gastrointestinal tract
* Antiosteoporotic drug
* Long term steroid treatment (within the last 12 months)
* Pregnancy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Serum concentration of C-terminal telopeptide (CTX) | -10 to 240 minutes
  Marker of bone resorption, measured in serum
N-terminal propeptide of type 1 procollagen (P1NP) | -10 to 240 minutes
  Marker of bone formation, concentration measured in serum

SECONDARY OUTCOMES:
PTH | -10 to 240 minutes
  PTH concentration measured in serum
Glucose-dependent insulinotropic polypeptide (GIP) | -10 to 240 minutes
  Gut hormone, concentration measured in plasma
Glucagon-like peptide-2 (GLP-2) | -10 to 240 minutes
  Gut hormone, concentration measured in plasma
Glucagon-like peptide-1 (GLP-1) | -10 to 240 minutes
  Gut hormone, concentration measured in plasma
Glucose | -10 to 240 minutes
  Glucose concentration measured in serum
Insulin | -10 to 240 minutes
  Insulin concentration measured in serum
C-peptide | -10 to 240 minutes
  C-peptide concentration measured in serum

OTHER OUTCOMES:
Blood pressure | -10 to 240 minutes
  Blood pressure (systolic and diastolic) measured before blood sampling
Heart rate | -10 to 240 minutes
  Heart rate measured before blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Mette Rosenkilde, MD, Study Director — University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided